CLINICAL TRIAL: NCT06640452
Title: RECOVERYFUN: An Integrated VR-based Tele-rehabilitation Platform to Support RECOVERY and Maintenance of FUNctional Abilities Among Seniors
Acronym: RECOVERYFUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government); European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_004_2024
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Home-based Rehabilitation; Older People
Keywords: app; virtual reality; technology-integrated rehabilitation; tele-rehabilitation platform
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- older adults (Experimental): The population concerned of patients who has overcome an acute event and completed intensive inpatient rehabilitation. The patient we are referring to has already returned home and needed to maintain the goals achieved or increase functionality.
  Interventions: Other: RecoveryFun system

INTERVENTIONS:
Other: RecoveryFun system — The system components were: VR headset; wereable biosensors, clinical platform, caregiver app and smart services.

SUMMARY:
The scope of the RecoveryFun study is to test a new personalised home rehabilitation solution to leverage the telehealth paradigm and increase the possibility for seniors to perform remotely supervised home-rehabilitation.

DETAILED DESCRIPTION:
This study was designed to test the usability and acceptability of the RecoveryFun system by a group of subjects, aged 60 years or older, within one year after an acute event with upper limb hemiplegia (Fugl- Meyer > 33). The patient, once the acute and intensive phase of rehabilitation is over, should also continue from home the process begun. However, this often creates difficulties for the patient. The study was carried out at the three recruitment sites (ZURZACH Care, TRAINM and INRCA)

The study was structured in two phases:

* A pilot in protected environment;
* A trial with the system used at the patient's home. The inclusion/exclusion criteria for the two steps were the same and the tools used to evaluate the result were the same too.

The two phases had different specific objectives and to avoid any bias due to previous experience the participants recruited in the two phases were different.

The RecoveryFun system comprehended Three tools: a Virtual reality headset for rehabilitation purposes, a set of Exergames and an app installed on caregiver's smartphone to motivate and support the end user in the therapy. The clinical personnel had access to the Clinical platform provided as a secured web app. The system administrator could differentiate access rights to each clinical user group (e.g: doctors, physiotherapists, nurses). An Innovative biosensing wireless sensor (wristband) was integrated in the connected ecosystem to measure physiological parameters (Heart Rate and Electrodermal Activity) of end users during the rehabilitation session. The patient performed the rehabilitation session according to the rehabilitation plan defined by the clinician. To have coherent results the rehabilitation plan included at least two weekly rehabilitation sessions lasting between 10 and 30 minutes, with the support of the caregiver, if necessary. Each session was planned and scheduled by the therapist remotely via the dedicated clinical platform.

After 4 weeks the assessment of usability and acceptability of the RecoveryFun system were performed by validated tools.

ELIGIBILITY:
Inclusion Criteria:

* No more than 12 months from acute event (for example stroke or brain injury)
* Trunk Impairment Scale (TIS) ≥20
* Fugl-Meyer Assessment Upper Extremities: Motor function for upper extremities (section A-D): a minimum Score of ≥33 is requested.

Exclusion Criteria:

* Technical Requirements based on the safety manual of the "Pico" headset
* Presence of pathology that could impact on the ability of using VR system or can be worsened by the use of VR system
* Montreal Cognitive Assessment (MoCA) score <24

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Usability of the RecoveryFun system | after 4 weeks of home-rehabilitation with RecoveryFun system
  The usability was assessed by the System Usability Scale (SUS). The SUS is a 10 item questionnaire with 5 response options.It generates a quantifiable measure called the SUS score, which ranges from 0 to 100, with zero being the least and 100 being the maximum.
Acceptability of the RecoveryFun system | after 4 weeks of home-rehabilitation with RecoveryFun system
  The acceptability was assessed by the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST). The QUEST is a 12-item outcome measure that assesses user satisfaction with two components, Device and Services. The questionnaire consists of 12 satisfaction items.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

REFERENCES:
- [Derived] Benadduci M, Franceschetti C, Marziali RA, Frese S, Sandor PS, Tombolesi V, Bozzi V, Rossi L. An Integrated Virtual Reality-Based Telerehabilitation Platform to Support Recovery and Maintenance of Functional Abilities Among Older Adults: Protocol for a Usability and Acceptability Study. JMIR Res Protoc. 2025 Jul 29;14:e68358. doi: 10.2196/68358. PMID 40729692